CLINICAL TRIAL: NCT06609252
Title: The Effect of Breast Milk Odour and Mother's Voice on Pain and Comfort During Retinopathy Examination in Premature Infants
Brief Title: Breast Milk Odour and Mother's Voice on Pain and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Atiye Karakul, Assoc. Prof., Tarsus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/74
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Pain; Breast Milk Odour; Comfort
Keywords: pain; breast milk odour; comfort
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- breast milk smell (Experimental): On the day of the study, the mothers of the babies will be contacted and fresh breast milk will be obtained from the mother of each baby. In the study, a sterile sponge will be used to smell the breast milk to the baby. Breast milk will be taken as 2 ml, dripped onto a sterile sponge and held 10 cm away from the baby's nose and sniffed 2 minutes before the examination.
  Interventions: Other: Breast milk odour
- mother's voice (Experimental): Mothers of premature babies in the mother voice group will be given a voice recorder on the day of the study and will be encouraged to express their feelings and thoughts and say what they want to say to their babies and will be asked to talk to their babies as they wish. The mother's voice, which is recorded 2 minutes before the procedure, will be placed approximately 30 cm away from the baby's ear and a loudspeaker will be placed at the foot end so that the baby can listen to the sound. The American Academy of Paediatrics recommends a sound level of 45-50 dB for premature babies. Therefore, the sound level will be measured with a decibel meter and set to 50 dB.
  Interventions: Other: Mother voice
- control (No Intervention): In the guideline prepared jointly by the Turkish Neonatology Association and the Turkish Society of Ophthalmology in 2021, it is recommended that the baby should be held by a nurse in such a way that the baby's head and arms are fixed, and the baby's hands and feet should be gently flexed or loosely swaddled during the retinopathy examination. Within the routine practice of the clinic, the babies in the control group are held.

INTERVENTIONS:
Other: Breast milk odour — On the day of the study, the mothers of the babies will be contacted and fresh breast milk will be obtained from the mother of each baby. In the study, a sterile sponge will be used to smell the breast milk to the baby. Breast milk will be taken as 2 ml, dripped onto a sterile sponge and held 10 cm away from the baby's nose and sniffed 2 minutes before the examination.
  Arms: breast milk smell
Other: Mother voice — Mothers of premature babies in the mother voice group will be given a voice recorder on the day of the study and will be encouraged to express their feelings and thoughts and say what they want to say to their babies and will be asked to talk to their babies as they wish. The mother's voice, which is recorded 2 minutes before the procedure, will be placed approximately 30 cm away from the baby's ear and a loudspeaker will be placed at the foot end so that the baby can listen to the sound.
  Arms: mother's voice

SUMMARY:
This study will be conducted to examine the effect of breast milk smell and mother's voice on pain and comfort in retinopathy examination in premature infants. The sample of the study will consist of premature infants who are receiving treatment and care in Izmir Provincial Health Directorate Izmir City Hospital Neonatal Intensive Care Unit within the central borders of Izmir province and who comply with the research limitations to be examined for ROP.

Stage 1: The research will start after the ethics committee and institutional permissions are obtained. The group in which the babies will be included will be determined by randomisation method. In the clinic where the research is carried out, ROP examination is performed on a certain day of the week, so the families of premature babies who meet the inclusion criteria will be informed about the research and their verbal and written permissions will be obtained.

Stage 2: On the day of the examination, fresh breast milk will be obtained from the mothers of the babies in the breast milk group. Mothers of premature infants in the mother voice group will be asked to make a voice recording before the examination. 'Introductory Information Form' will be filled out before the procedure.

Stage 3: Video recording will be made to evaluate the pain, stress, comfort and physiological parameters of premature babies. Video recording will be started 2 minutes before the examination. Video recording will continue for 5 minutes after the ROP examination.

Stage 4: Breast milk odour, mother's voice and physiological parameters of the babies in the control group will be recorded 2 minutes before the examination, 2 minutes after the end of the examination and 5 minutes after the end of the examination.

Stage 5: The babies in the breast milk odour group will be made to smell the styrene sponge dripped with their own mother's milk 2 minutes before the procedure.

Stage 6: Babies in the mother's voice group will be made to listen to their own mother's voice 2 minutes before the procedure.

7th Stage: Babies in the control group will be subjected to the routine practice of the clinic.

Stage 8: The videos recorded after the interventions and the scores given to the PIPP, CEQ, and PBQ scales will be evaluated by two independent faculty members who are experts in their fields.

DETAILED DESCRIPTION:
The use of effective and efficient non-pharmacological methods to reduce the pain and stress experienced by premature babies due to retinopathy examination and to increase their comfort has an important place in supporting optimal growth and development. This study was planned to reveal the effectiveness of different non-pharmacological methods during the examination performed within the scope of the screening programme for prematurity.

This study will be conducted to examine the effect of breast milk smell and mother's voice on pain and comfort in retinopathy examination in premature infants. The sample of the study will consist of premature infants who are receiving treatment and care in Izmir Provincial Health Directorate Izmir City Hospital Neonatal Intensive Care Unit within the central borders of Izmir province and who comply with the research limitations to be examined for ROP.

Data Collection Breast milk odour group: On the day of the study, the mothers of the babies will be contacted and fresh breast milk will be obtained from the mother of each baby. In the study, a sterile sponge will be used to smell the breast milk to the baby. Breast milk will be taken as 2 ml, dripped onto a sterile sponge and held 10 cm away from the baby's nose and sniffed 2 minutes before the examination.

Mother voice group: Mothers of premature babies in the mother voice group will be given a voice recorder on the day of the study and will be encouraged to express their feelings and thoughts and say what they want to say to their babies and will be asked to talk to their babies as they wish. The mother's voice, which is recorded 2 minutes before the procedure, will be placed approximately 30 cm away from the baby's ear and a loudspeaker will be placed at the foot end so that the baby can listen to the sound. The American Academy of Paediatrics recommends a sound level of 45-50 dB for premature babies. Therefore, the sound level will be measured with a decibel meter and set to 50 dB.

Control group: In the guideline prepared jointly by the Turkish Neonatology Association and the Turkish Society of Ophthalmology in 2021, it is recommended that the baby should be held by a nurse in such a way that the baby's head and arms are fixed, and the baby's hands and feet should be gently flexed or loosely swaddled during the retinopathy examination. Within the routine practice of the clinic, the babies in the control group are held.

Stage 1: The research will start after the ethics committee and institutional permissions are obtained. The group in which the babies will be included will be determined by randomisation method. In the clinic where the research is carried out, ROP examination is performed on a certain day of the week, so the families of premature babies who meet the inclusion criteria will be informed about the research and their verbal and written permissions will be obtained.

Stage 2: On the day of the examination, fresh breast milk will be obtained from the mothers of the babies in the breast milk group. Mothers of premature infants in the mother voice group will be asked to make a voice recording before the examination. 'Introductory Information Form' will be filled out before the procedure.

Stage 3: Video recording will be made to evaluate the pain, stress, comfort and physiological parameters of premature babies. Video recording will be started 2 minutes before the examination. Video recording will continue for 5 minutes after the ROP examination.

Stage 4: Breast milk odour, mother's voice and physiological parameters of the babies in the control group will be recorded 2 minutes before the examination, 2 minutes after the end of the examination and 5 minutes after the end of the examination.

Stage 5: The babies in the breast milk odour group will be made to smell the styrene sponge dripped with their own mother's milk 2 minutes before the procedure.

Stage 6: Babies in the mother's voice group will be made to listen to their own mother's voice 2 minutes before the procedure.

7th Stage: Babies in the control group will be subjected to the routine practice of the clinic.

Stage 8: The videos recorded after the interventions and the scores given to the PIPP, CEQ, and PBQ scales will be evaluated by two independent faculty members who are experts in their fields.

ELIGIBILITY:
Inclusion Criteria:

* Parent's infant agreeing to participate in the study
* The baby is being treated and monitored in the Neonatal Intensive Care Unit
* The mother has milk
* Gestational age ≤32 weeks
* Birth weight ≤2000 grams
* Babies who will be examined for ROP for the first time

Exclusion Criteria:

* Gestational age of 33> weeks
* No need for mechanical ventilator support,
* Hearing sensory loss diagnosis
* Administration of sedative, analgesic and anticonvulsant drugs before the examination
* Having a neurological problem (e.g. asphyxia, hypoxic ischaemic encephalopathy, intraventricular

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
pain level | 1 hour
  Premature Newborn Pain Profile It is a pain diagnostic scale developed by Stevens et al. It was revised by Gibbins et al. for premature infants at 26-37 gestation weeks. Turkish validity and reliability was performed by Akcan and Yiğit in 2015. Statements including 7 items such as gestational age, behavioural status, highest heart rate value, lowest oxygen saturation value, forehead wrinkling, squinting and widening of the wings of the nose are questioned. Each item is scored as 0, 1, 2, 3 from good to bad. The baby's pain is calculated over the total score. The highest score is 21 and the lowest score is 0. If the pain is mild, it is evaluated by scoring between 0-6 points, moderate severity between 7-12 points, and severe between 13-21 points.
stress level | 1 hour
  Neonatal Stress Scale It was developed by Ceylan and Bolışık to evaluate stress in premature infants and its validity and reliability were performed. The scale is a three-point Likert-type scale and consists of 24 items and 8 sub-dimensions. The scale consists of 'facial expression', 'body colour', 'respiration', 'activity level', 'comfortability', 'muscle tone', 'excursions' and 'posture' sub-dimensions. Each subgroup in the scale is scored between 0-2 points. The minimum score that can be obtained from the scale is 0 and the maximum score is 16. An increase in the score indicates an increase in the infant's stress. The evaluation of the scale is done through observation
comfort level | 1 hour
  Premature Infant Comfort Scale Alemdar and Tüfekçi adapted this scale, which was developed by Caljouw et al. in 2007 for premature infants, into Turkish and stated that it evaluates 7 parameters such as 'Alertness, Calmness / Agitation, Respiratory Status (only in mechanical ventilation support) or Crying (not evaluated because it was scored only in children with spontaneous breathing), Physical Movement, Muscle Tone, Facial Movements and Mean Heart Rate.' Each condition is scored from 1 to 5, ranging from good to bad, with 35 being the lowest and 7 being the highest comfort score.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Tarsus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yue W, Han X, Luo J, Zeng Z, Yang M. Effect of music therapy on preterm infants in neonatal intensive care unit: Systematic review and meta-analysis of randomized controlled trials. J Adv Nurs. 2021 Feb;77(2):635-652. doi: 10.1111/jan.14630. Epub 2020 Nov 17. PMID 33200833
- [Background] Fajolu IB, Dedeke IOF, Ezenwa BN, Ezeaka VC. Non-pharmacological pain relief interventions in preterm neonates undergoing screening for retinopathy of prematurity: a systematic review. BMJ Open Ophthalmol. 2023 Dec 6;8(1):e001271. doi: 10.1136/bmjophth-2023-001271. PMID 38057104
- [Background] Valeri BO, Holsti L, Linhares MB. Neonatal pain and developmental outcomes in children born preterm: a systematic review. Clin J Pain. 2015 Apr;31(4):355-62. doi: 10.1097/AJP.0000000000000114. PMID 24866853
- [Background] Asadollahi M, Jabraeili M, Mahallei M, Asgari Jafarabadi M, Ebrahimi S. Effects of Gentle Human Touch and Field Massage on Urine Cortisol Level in Premature Infants: A Randomized, Controlled Clinical Trial. J Caring Sci. 2016 Sep 1;5(3):187-194. doi: 10.15171/jcs.2016.020. eCollection 2016 Sep. PMID 27752484
- [Background] Dilli D, Ilarslan NE, Kabatas EU, Zenciroglu A, Simsek Y, Okumus N. Oral sucrose and non-nutritive sucking goes some way to reducing pain during retinopathy of prematurity eye examinations. Acta Paediatr. 2014 Feb;103(2):e76-9. doi: 10.1111/apa.12454. Epub 2013 Nov 11. PMID 24730361
- [Background] Jang EK, Lee H, Jo KS, Lee SM, Seo HJ, Huh EJ. Comparison of the Pain-relieving Effects of Human Milk, Sucrose, and Distilled Water during Examinations for Retinopathy of Prematurity: A Randomized Controlled Trial. Child Health Nurs Res. 2019 Jul;25(3):255-261. doi: 10.4094/chnr.2019.25.3.255. Epub 2019 Jul 31. PMID 35004418
- [Background] Liao, W. H., Xu, H. Y., Zhou, X., Tian, J. L., Fang, X. Y., Ding, J., … Wu, H. L. (2019). Non-nutritive sucking and nesting greatly reduces pain during retinopathy screening in premature infants. Hong Kong Journal of Paediatrics, 24(3).